CLINICAL TRIAL: NCT01766869
Title: Improving Cancer Foci Detection in Prostate Cancer Using Multiparametric MRI/MRS and Machine Learning to Better Manage the Disease
Brief Title: Improving Cancer Foci Detection in Prostate Cancer Using Multiparametric MRI/MRS
Acronym: GCC 1261
Status: Withdrawn | Type: Observational
Why Stopped: No participants enrolled
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Principal Investigator, University of Maryland, Baltimore
Other Study IDs: HP-00054431
Record Dates: First submitted 2013-01-08; First posted 2013-01-11 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; MRI/MRS
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigators' goal is to develop a non-selective and non-invasive procedure to identify aggressive tumors and simultaneously identify their exact location in Prostate cancer patients undergoing radical prostatectomy by combining multiparametric MRI and machine learning techniques. The combination of multi-parametric MRI and machine learning (validated using histopathology) can lead to increased sensitivity and specificity of cancer foci in the prostate, and help in isolating aggressive from indolent tumors. This increased sensitivity and specificity may eventually lead to: a) a reduction in the number of patients that undergo unnecessary treatment, and b) enhance current treatment options by enabling the use of focused therapies. The investigators will recruit 15 patients with prostate cancer that are currently scheduled to undergo radical prostatectomy into the study. All patients will obtain an advanced MRI study prior to the radical prostatectomy. MRI scans will include a) high-resolution volumetric images using T1 and T2-weighted imaging, b) vascular images using dynamic contrast enhanced (DCE) imaging, c) biophysical microstructure images using diffusion-weighted imaging, and d) biochemical images using MR spectroscopic imaging. Following radical prostatectomy, a pathologist will grade the prostatectomy specimens based on standard of care (Gleason grading system). Correlations will be generated between the parameters obtained from scans and from clinical assessments.

ELIGIBILITY:
Inclusion Criteria:

1. All male patients that have opted for radical prostatectomy
2. Subjects must be capable of giving informed consent.
3. Subjects must not be claustrophobic.

Exclusion Criteria:

1. Subjects with pacemakers.
2. Subjects who have metallic ferromagnetic implants or pumps.
3. All females are excluded from this study.
4. Subjects with kidney disease of any severity or on hemodialysis.
5. Subjects with known allergies to gadolinium-based contrast agents.
6. Subjects incapable of lying on their backs for up to an hour at a time.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: prostate cancer patients that have elected to go for radical prostatectomy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Primary Objective: distinguishing high-grade tumors vs. low-grade tumors and normal prostate | 16 months
  Whether advanced MR imaging techniques can be used to train machine-learning techniques to distinguish high-grade tumors from low-grade tumors and normal prostate. The machine-learning techniques will be trained using histopathology data as the ground truth.
  To achieve this we will obtain volumetric images of the various tissue attributes (listed below) and match them to histopathology:
  * Vascular permeability (ktrans) using dynamic contrast enhanced MRI (DCE-MRI)
  * Morphological changes captured using T2 and diffusion changes using diffusion weighted MRI (DW-MRI)
  * Metabolic signatures of (choline+creatine)/citrate) or CC/C using magnetic resonance spectroscopic imaging (MRSI)
  * Correlate in vivo imaging findings to ex vivo histopathology using deformable image registration
  * Develop a multiclass support vector machine (SVM) using the set of multi-parametric images as input, and use it predict a score akin to the Gleason score.

SECONDARY OUTCOMES:
Secondary Objective: non-invasive and quantitative test to accurately identify the tumor grade and location. | 16 months
  Advanced MR imaging techniques can be used alone in classifying tumor grade. Datasets collected will be partitioned into subsets that will be used for testing the machine learning techniques. For example: 90% of the data will be used for training and the remaining 10% will be used for testing. This process will be repeated over a combination of different subsets. Our hypothesis is that Machine Learning methods will assist in analyzing the differences between aggressive tumors, indolent tumors, and normal tissue. We further hypothesize this analysis will help in synthesizing an imaging-based "score" that can identify an aggressive tumor from indolent tumors and normal tissue in new cases after training. We believe using multi-parametric MRI combined with an advanced machine learning technique can improve the sensitivity and specificity of tumor foci detection. This will result in a non-invasive and quantitative test to accurately identify the tumor grade and location.

CONTACTS AND LOCATIONS:
Overall Officials: Warren D'Souza, PhD, Principal Investigator — UMD
Locations (1):
- Ummc Msgcc, Baltimore, Maryland, United States